CLINICAL TRIAL: NCT03862274
Title: Examining Developmental Outcomes of Children Diagnosed With CLN2 Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Jessica Scherr (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Jessica Scherr, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB18-00464
Record Dates: First submitted 2019-01-04; First posted 2019-03-05 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Batten Disease; CLN2; Neuronal Ceroid-Lipofuscinoses
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CLN2 Natural History Control Group: Patients that have a TPP1 enzyme deficiency and/or confirmed molecular diagnosis of pathogenic variants in the TPP1 gene are eligible to participate if they are untreated or not receiving cerliponase alfa.
- CLN2 Treatment Group: Patients that have a TPP1 enzyme deficiency and/or confirmed molecular diagnosis of pathogenic variants in the TPP1 gene are eligible to participate if they are receiving cerliponase alfa.
  Interventions: Other: CLN2 Treatment

INTERVENTIONS:
Other: CLN2 Treatment — Patients that have a TPP1 enzyme deficiency and/or confirmed molecular diagnosis of pathogenic variants in the TPP1 gene are eligible to participate if they are receiving cerliponase alfa.
  Groups: CLN2 Treatment Group

SUMMARY:
The investigators propose a study to assess cognitive and developmental outcomes of patients with CLN2 that are untreated and receiving cerliponase alfa. This study aims to validate standardized assessment measures to establish a standard of care. The secondary aim is to compare cognitive and developmental outcomes of patients with CLN2 that are receiving celiponase alfa to a natural history cohort. To accomplish specific aims of the study, the investigators will use a multi-method approach to collect retrospective data collected as standard of care and prospective developmental data in children with CLN2 disease. The investigators will use a combination of standardized measures that include direct assessment and parent report of child development. The investigators focus will also include multiple measures of development including language, motor, social-emotional, and adaptive functioning.

DETAILED DESCRIPTION:
CLN2 disease is a predominantly late infantile form of neuronal ceroid lipofuscinosis and one of the many genetic isoforms of Batten disease. Mutations in the CLN2 gene are characterized by deficient lysosomal serine protease TPP1, an enzyme that metabolizes intracellular lysosomal storage materials. Accumulations of intracellular deposits occur over time and in many organs of individuals with CLN2 disease and lead to neurodegeneration and, eventually, death. CLN2 disease is an extremely rare genetic disease affecting around 1 per 200,000 live births. Symptoms emerge early in life typically between the ages of 2 and 4 years of age and include seizures, as well as loss of motor, language, and vision functioning. Development further declines in early childhood and by age 6 years, children with CLN2 are often unable to walk or sit unsupported and become blind. The progression of the disease is rapid with death typically occurring in mid-childhood between the ages of 10 and 15 years of age.

Recently, enzyme replacement therapy (ERT), cerliponase alfa, which is a recombinant form of human TPPI, was the first FDA-approved treatment to slow the progression of motor decline in children with CLN2. Cerliponase alfa is expected to restore TPP1 enzyme activity in the brain and alter neurodegeneration and disease progression. Animal models suggest promising treatment outcomes as cerliponase alfa significantly delayed the onset of clinical signs, preserved motor and cognitive function, and prolonged life. Initial results from a clinical trial further demonstrated that patients receiving cerliponase alfa had less motor declines, as measured by the CLN2 Clinical Rating Scale, compared to a natural history cohort. Despite these promising results, little is known about the trajectory of other developmental domains, including language, social-emotional, and adaptive functioning of children receiving cerliponase alfa. Likewise, the developmental trajectory of untreated patients with CLN2 is not well understood. Therefore, it is important to understand developmental outcomes and the progression of CLN2 in a natural history cohort in order to compare the effectiveness of treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have a TPP1 enzyme deficiency
* Patients have confirmed molecular diagnosis of pathogenic variants in the TPP1 gene
* Patients that are enrolled in post-marketing studies will be allowed to enroll into the current study

Exclusion Criteria:

* Patients without a diagnosis of CLN2 and deficiency of TPP1
* Patients that are currently enrolled as part of a larger multi-center clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have a TPP1 enzyme deficiency and/or confirmed molecular diagnosis of pathogenic variants in the TPP1 gene are eligible to participate if they are untreated or are receiving cerliponase alfa.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Visual Reception Skills on the Mullen Scales of Early Learning | up to 4 years
  Changes in the Visual Reception subscale on the Mullen Scales of Early Learning will be assessed every 6 months. Visual reception skills are a measure of visual processing and problem solving. Raw scores will be used as a measure of visual receptions skills with scores ranging from 0 to 50. Higher scores indicate more visual reception skills.
Changes in Fine Motor Skills on the Mullen Scales of Early Learning | up to 4 years
  Changes in the Fine Motor subscale on the Mullen Scales of Early Learning will be assessed every 6 months. Fine motor skills are a measure of fine motor coordination. Raw scores will be used as a measure of fine motor skills with scores ranging from 0 to 49. Higher scores indicate more fine motor skills.
Changes in Receptive Language Skills on the Mullen Scales of Early Learning | up to 4 years
  Changes in the Receptive Language subscale on the Mullen Scales of Early Learning will be assessed every 6 months. Receptive language skills are a measure of the understanding of language. Raw scores will be used as a measure of receptive language skills with scores ranging from 0 to 48. Higher scores indicate more receptive language skills.
Changes in Expressive Language Skills on the Mullen Scales of Early Learning | up to 4 years
  Changes in the Expressive Language subscale on the Mullen Scales of Early Learning will be assessed every 6 months. Expressive language skills are a measure of how an individual communicates. Raw scores will be used as a measure of expressive language skills with scores ranging from 0 to 50. Higher scores indicate more expressive language skills.
Motor and Language Changes on the CLN2 disease rating scale | up to 4 years
  Change in motor and language subscales of the CLN2 disease rating scale. Ranges for scores are 0 to 6 with higher scores indicating more abilities in motor and language skill development.

SECONDARY OUTCOMES:
Changes in Receptive Language Skills on the Preschool Language Scales | up to 4 years
  Changes in the Receptive Language subscale on the Preschool Language Scales will be assessed every 6 months. Receptive language skills are a measure of the understanding of language. Raw scores will be used as a measure of receptive language skills with scores ranging from 0 to 65. Higher scores indicate more receptive language skills.
Changes in Expressive Language Skills on the Preschool Language Scales | up to 4 years
  Changes in the Expressive Language subscale on the Preschool Language Scales will be assessed every 6 months. Expressive language skills are a measure of how an individual communicates. Raw scores will be used as a measure of expressive language skills with scores ranging from 0 to 67. Higher scores indicate more expressive language skills.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scherr, PhD, Principal Investigator — Nationwide Children's Hospital; Emily de los Reyes, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulz A, Kohlschutter A, Mink J, Simonati A, Williams R. NCL diseases - clinical perspectives. Biochim Biophys Acta. 2013 Nov;1832(11):1801-6. doi: 10.1016/j.bbadis.2013.04.008. Epub 2013 Apr 17. PMID 23602993
- [Background] Schulz A, Ajayi T, Specchio N, de Los Reyes E, Gissen P, Ballon D, Dyke JP, Cahan H, Slasor P, Jacoby D, Kohlschutter A; CLN2 Study Group. Study of Intraventricular Cerliponase Alfa for CLN2 Disease. N Engl J Med. 2018 May 17;378(20):1898-1907. doi: 10.1056/NEJMoa1712649. Epub 2018 Apr 24. PMID 29688815
- [Background] Wisniewski KE, Zhong N, Philippart M. Pheno/genotypic correlations of neuronal ceroid lipofuscinoses. Neurology. 2001 Aug 28;57(4):576-81. doi: 10.1212/wnl.57.4.576. PMID 11548735
- [Background] Worgall S, Kekatpure MV, Heier L, Ballon D, Dyke JP, Shungu D, Mao X, Kosofsky B, Kaplitt MG, Souweidane MM, Sondhi D, Hackett NR, Hollmann C, Crystal RG. Neurological deterioration in late infantile neuronal ceroid lipofuscinosis. Neurology. 2007 Aug 7;69(6):521-35. doi: 10.1212/01.wnl.0000267885.47092.40. PMID 17679671
- [Background] Williams RE, Aberg L, Autti T, Goebel HH, Kohlschutter A, Lonnqvist T. Diagnosis of the neuronal ceroid lipofuscinoses: an update. Biochim Biophys Acta. 2006 Oct;1762(10):865-72. doi: 10.1016/j.bbadis.2006.07.001. Epub 2006 Jul 12. PMID 16930952